CLINICAL TRIAL: NCT00587132
Title: Pilot Study Using Secretin and Iodinated Intravenous Contrast and 64-Channel CT in Patients at High Risk for Pancreatic Adenocarcinoma
Brief Title: Secretin (ChiRhoStim) Pancreas Perfusion for Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Collaborators: ChiRhoClin, Inc. (Industry)
Responsible Party: Principal Investigator, Naoki Takahashi, Associate Professor of Radiology,College of Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 231-06
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2013-06-20 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Pancreatic Cancer
Keywords: Diabetes mellitus; Peutz-Jeghers syndrome
MeSH Terms: conditions — Pancreatic Neoplasms; Diabetes Mellitus; Peutz-Jeghers Syndrome | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- New Onset Diabetes (Experimental): Adults diagnosed diabetes within two years, and at least one of the following: no family history of diabetes, abdominal discomfort, anorexia, weight loss, elevated serum cancer antigen 19-9 (CA 19-9), or those undergoing endoscopic ultrasound (EUS) with or without Fine Needle Aspiration (FNA) for pancreatic cancer screening.
  All subjects on this arm will receive Synthetic Human Secretin as a 0.2mcg/kg one time dose prior to CT imaging on Day 1 of the study.
  Interventions: Drug: Synthetic Human Secretin
- Familial Pancreatic Cancer (Experimental): Adults age 35-99 with familial pancreatic cancer with two or more first degree relatives with pancreatic cancer.
  All subjects on this arm will receive Synthetic Human Secretin as a 0.2mcg/kg one time dose prior to CT imaging on Day 1 of the study.
  Interventions: Drug: Synthetic Human Secretin
- Peutz-Jeghers Syndrome (Experimental): Adults age 35-99 with Peutz-Jeghers syndrome.
  All subjects on this arm will receive Synthetic Human Secretin as a 0.2mcg/kg one time dose prior to CT imaging on Day 1 of the study.
  Interventions: Drug: Synthetic Human Secretin
- Clinical Symptoms of Pancreatic Cancer, Normal CT (Experimental): Adults age 35-99 with suspicious clinical symptoms of pancreatic cancer, but had normal CT of the abdomen with iodinated contrast within 2 weeks.
  All subjects on this arm will receive Synthetic Human Secretin as a 0.2mcg/kg one time dose prior to CT imaging on Day 1 of the study.
  Interventions: Drug: Synthetic Human Secretin

INTERVENTIONS:
Drug: Synthetic Human Secretin — 0.2mcg/kg one time dose.
  Other Names: ChiRhoStim

SUMMARY:
The purpose of this study is to test if secretin-enhanced CT is a useful noninvasive screening tool for pancreatic cancer in a high-risk population.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth most common cause of cancer death in the US. Because patients with pancreatic cancer rarely presents with disease specific symptoms until late in the course of the disease, identifying and developing surveillance strategies for early detection of asymptomatic pancreatic cancer is critical. EUS and fine needle aspirate (FNA) are currently the most accurate non-operative methods of establishing the presence or absence of pancreatic cancer.

The CT findings of pancreatic cancer include an attenuation difference between the pancreatic mass and the surrounding pancreatic parenchyma, pancreatic ductal dilation and cutoff, disruption of the normal fatty marbling of the pancreatic parenchyma, rounding of the inferior margin of the posterior head of the pancreas, atrophy of the proximal gland, and signs of locally advanced or distant disease. In a case-controlled retrospective review of pancreatic cancers missed at CT prior to clinical presentation at the Mayo Clinic, Gangi et al found that CT findings definite or suspicious for pancreatic cancer were present in 50% of scans obtained up to 18 months before the clinical diagnosis of pancreatic cancer. Pancreatic duct dilation and cutoff were early CT findings indicating tumor presence, and were associated with near-perfect and substantial interobserver agreement. Consequently, early pancreatic neoplasms likely result in at least partial occlusion of the duct, leading to subsequent ductal dilation.

We hypothesize that increased production of the pancreatic juice distends the otherwise small caliber pancreatic duct, and accentuate the secondary sign of pancreatic duct obstruction by a small pancreatic mass. The investigators will be able to take advantage of this physiologic effect of secretin, by obtaining multi-planar scans with isotropic resolution using a 64-channel CT system.

Secretin is a safe agent that increases pancreatic exocrine secretion. Intravenously administered secretin increases the pancreatic juice secretion, and magnetic resonance or CT scan obtained after secretin has been shown to improve visualization of the pancreatic duct.

Day 1: Patient will fast 4 hours prior to the study. 1 L of water is given by mouth as an oral contrast material 30 minutes prior to the study. After placing an angiocath in the antecubital fossa, the patient will be placed in a supine position on the CT scanner.

Secretin test dose will be given intravenously (0.2mcg (0.1ml). If no reaction is noted after one minute, then Secretin will be given intravenously (0.2 mcg/kg IV slowly over one minute). If an allergic reaction is noted, the patient will not have a CT scan performed as part of this study protocol, and that participant will be ineligible to participant with this study. Secretin bolus will be terminated if Systolic BP < 90mm/Hg is not corrected with IV fluids.

Pre-contrast scan will be obtained with collimation of 0.6 x 64 mm and a pitch of 1.2 through the abdomen under deep inspiration. Images will be reconstructed with 1 mm slice thickness and 2 mm increment.

Five minutes after administration of the intravenous Secretin, iodinated contrasted Omnipaque 350 administered at 3-5ml/sec. Post-iodine-contrast scanning will be obtained with collimation of 0.6 x 64 mm and a pitch of 1.2 through the abdomen with scan delays of 40- and 70-seconds. Total of 150 ml of intravenous iodinated contrast will be administered at the rate of 3 - 5 ml/ sec.

For the 3 month (Day 2) and 18 month (Day 3) follow-up CT imaging:

Patient will fast four hours before scan. 1 liter of water given orally 30 minutes prior to scan. An IV will be placed, and participant will have iodinated contrast (Omnipaque 350) administered at 3-5ml/sec. Post iodine scanning will be done with collimation of 0.6 x64mm and a pitch of 1.2 through the abdomen with scan delays of 40 and 70 seconds.

For the optional CT scan for those who have initial positive CT:

This exam is to be done only before endoscopic ultrasound (EUS). Patient will fast four hours before scan. 1 liter of water given orally 30 minutes prior to scan. An IV will be placed, and participant will have iodinated contrast (Omnipaque 350) administered at 3-5ml/sec. Post iodine scanning will be done with collimation of 0.6 x64mm and a pitch of 1.2 through the abdomen with scan delays of 40 and 70 seconds.

Subjects will be followed up for 3-5 years to determine if they develop pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Persons 50 years or older with recently diagnosed diabetes (within 2 years), with at least one of the following: no family history of diabetes, abdominal discomfort, anorexia, weight loss, elevated serum CA 19-9, or those undergoing EUS with or without Fine Needle Aspiration (FNA) for pancreatic cancer screening ; OR
* Persons 35 years old or older with familial pancreatic cancer with 2 or more first degree relatives with pancreatic cancer; OR
* Persons 35 years old or older with Peutz-Jeghers syndrome; OR
* Persons 35 years old or older with suspicious clinical symptoms of pancreatic cancer, but had normal CT of the abdomen with iodinated contrast within 2 weeks.

Exclusion Criteria:

* Persons with contraindication to iodinated contrast
* Allergy to iodinated contrast
* Renal insufficiency (serum creatinine > 1.5 mg/dl)
* Patients with contraindication to ionizing radiation
* Pregnancy
* Patients with previous pancreatic surgery
* Contraindication to secretin
* Allergy to secretin
* Acute pancreatitis

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Takahashi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mayo Clinic in Rochester, Minnesota from November 2006 until April 2009.
Groups:
- Familial Pancreatic Cancer: Adults age 35-99 with familial pancreatic cancer with two or more first degree relatives with pancreatic cancer
  All subjects on this arm will receive Synthetic Human Secretin as a 0.2mcg/kg one time dose prior to CT imaging on Day 1 of the study.
- Clinical Symptoms of Pancreatic Cancer, Normal CT: Adults age 35-99 with suspicious clinical symptoms of pancreatic cancer, but had normal CT of the abdomen with iodinated contrast within 2 weeks.
Period: Overall Study
Arm/Group | New Onset Diabetes | Familial Pancreatic Cancer | Peutz-Jeghers Syndrome | Clinical Symptoms of Pancreatic Cancer, Normal CT
Started | 4 | 0 | 0 | 0
Completed | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- New Onset Diabetes: 10 adults, diagnosed diabetes within two years, and at least one of the following: no family history of diabetes, abdominal discomfort, anorexia, weight loss, elevated serum cancer antigen 19-9 (CA 19-9), or those undergoing endoscopic ultrasound (EUS) with or without Fine Needle Aspiration (FNA) for pancreatic cancer screening.
  All subjects on this arm will receive Synthetic Human Secretin as a 0.2mcg/kg one time dose prior to CT imaging on Day 1 of the study.
- Familial Pancreatic Cancer: 10 adults age 35-99 with familial pancreatic cancer with two or more first degree relatives with pancreatic cancer
  All subjects on this arm will receive Synthetic Human Secretin as a 0.2mcg/kg one time dose prior to CT imaging on Day 1 of the study.
- Peutz-Jeghers Syndrome: 10 adults age 35-99 with Peutz-Jeghers syndrome.
  All subjects on this arm will receive Synthetic Human Secretin as a 0.2mcg/kg one time dose prior to CT imaging on Day 1 of the study.
- Clinical Symptoms of Pancreatic Cancer, Normal CT: 10 adults age 35-99 with suspicious clinical symptoms of pancreatic cancer, but had normal CT of the abdomen with iodinated contrast within 2 weeks.
- Total: Total of all reporting groups
Arm/Group | New Onset Diabetes | Familial Pancreatic Cancer | Peutz-Jeghers Syndrome | Clinical Symptoms of Pancreatic Cancer, Normal CT | Total
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 4
Age Categorical [Number; unit: participants]
  <=18 years | 0 |  |  |  | 0
  Between 18 and 65 years | 2 |  |  |  | 2
  >=65 years | 2 |  |  |  | 2
Gender [Number; unit: participants]
  Female | 3 |  |  |  | 3
  Male | 1 |  |  |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 |  |  |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Evidence of Pancreatic Tumor or Any Secondary Findings of Pancreatic Tumor as Shown by CT.
Description: Subjects will receive the secretin test dose just prior to the CT scan. Definitions: Evidence of Pancreatic Tumor (low-attenuation mass), Secondary Findings of Pancreatic Tumor such as dilated pancreatic duct or liver masses suggestive of liver metastases.
Time Frame: Day 1 of study
Population: All subjects had a normal CT scan. The study was terminated early due to lack of funding. No analysis was done due to the low enrollment.
Measure: Number; unit: participants
Groups:
- New Onset Diabetes: Adults, diagnosed diabetes within two years, and at least one of the following: no family history of diabetes, abdominal discomfort, anorexia, weight loss, elevated serum cancer antigen 19-9 (CA 19-9), or those undergoing endoscopic ultrasound (EUS) with or without Fine Needle Aspiration (FNA) for pancreatic cancer screening.
  All subjects on this arm will receive Synthetic Human Secretin as a 0.2mcg/kg one time dose prior to CT imaging on Day 1 of the study.
Arm/Group | New Onset Diabetes | Familial Pancreatic Cancer | Peutz-Jeghers Syndrome | Clinical Symptoms of Pancreatic Cancer, Normal CT
Number analyzed (Participants) | 4 | 0 | 0 | 0
participants | 0 |  |  |

ADVERSE EVENTS:
Arm/Group | New Onset Diabetes | Familial Pancreatic Cancer | Peutz-Jeghers Syndrome | Clinical Symptoms of Pancreatic Cancer, Normal CT
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No